CLINICAL TRIAL: NCT02702791
Title: Enhancing Physical Activity to Achieve Sustainable Benefits in Extrapulmonary Consequences of COPD
Brief Title: Sustaining Training Effects Through Physical Activity
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Thierry Troosters, Prof, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s57963
Record Dates: First submitted 2016-01-12; First posted 2016-03-09 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Physical activity; Pulmonary rehabilitation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Telecoaching - feasible goal setting and feedback to enhance patient's motivation and commitment - in addition to pulmonary rehabilitation.
  Interventions: Behavioral: Telecoaching; Other: pulmonary rehabilitation
- Usual care (Other): includes only general advices regarding physical activity.
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Telecoaching — Pedeometer based goals and telecoaching support
  Arms: Intervention
Other: pulmonary rehabilitation — Conventional pulmonary rehabilitation along the ATS-ERS guidelines, total duration 6 months.

SUMMARY:
This randomized control trial will investigate whether the implementation of a telecoaching program, initiated during pulmonary rehabilitation, is able to increase and maintain physical activity and general benefits until six months after rehabilitation discharge.

After three months of pulmonary rehabilitation (3 times a week), patients with COPD will be randomized to either an intervention group which receives an additional telecoaching program on top of the pulmonary rehabilitation, or to the usual care group, which only receives rehabilitation program. Apart from the added telecoaching program to the intervention group, the rehabilitation program will be identical and last for another three months (2 times a week). After discharge, both groups will be followed up for six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of COPD according to internationally accepted guidelines
* Patients that completed three months of the outpatient pulmonary rehabilitation program of Gasthuisberg University Hospital (Leuven, Belgium)
* Current or previous smoking exposure of at least 10 pack years
* Ability to manage electronic devices (smartphone, step counter)

Exclusion Criteria:

* Other predominant respiratory diseases than COPD (asthma, pulmonary hypertension)
* Orthopedic, neurological and muscular co morbidities that could interfere with normal biomechanical movement patterns and the ability to increase physical activity levels
* Patients on the waiting list for lung transplantation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Changes in physical activity (number of steps) | At three and six months of pulmonary rehabilitation and three and six months of follow up

SECONDARY OUTCOMES:
Changes in physical activity (time spent in moderate activity) | At three and six months of pulmonary rehabilitation and three and six months of follow up
Changes in pulmonary rehabilitation outcomes (Quadriceps force) | At three and six months of pulmonary rehabilitation and three and six months of follow up
Changes in pulmonary rehabilitation outcomes (Functional exercise capacity) | At three and six months of pulmonary rehabilitation and three and six months of follow up
Changes in pulmonary rehabilitation outcomes (Maximal exercise capacity) | At three and six months of pulmonary rehabilitation and six months of follow up
Changes in pulmonary rehabilitation outcomes (Endurance exercise capactity) | At three and six months of pulmonary rehabilitation and six months of follow up
Changes in pulmonary rehabilitation outcomes (Quality of life) | At three and six months of pulmonary rehabilitation and six months of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Troosters, PhD, Principal Investigator — Katholiek Universiteit Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Derived] Loeckx M, Rodrigues FM, Blondeel A, Everaerts S, Janssens W, Demeyer H, Troosters T. Sustaining training effects through physical activity coaching (STEP): a randomized controlled trial. Int J Behav Nutr Phys Act. 2023 Oct 10;20(1):121. doi: 10.1186/s12966-023-01519-w. PMID 37814266